CLINICAL TRIAL: NCT03108001
Title: Glowing and Expecting Follow Up
Status: Recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 206188
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Lean mothers: Participants that were in Glowing born from Lean mothers.
- Overweight mothers: Participants that were in Glowing born from Overweight mothers.
- Obese mothers: Participants that were in Glowing born from Obese mothers.
- Exercise group mothers: Participants that were in Expecting born from mothers that were in the exercise group.
- Non Exercise group mothers: Participants that were in Expecting born from mothers that were in the non- exercise group.

SUMMARY:
This study will help us learn more about how a mother's health during pregnancy may influence her child's growth and development later in life.

DETAILED DESCRIPTION:
This study will follow participants who participated in the Glowing and Expecting study. 514 people who are 5 to 14 years of age who agreed to be contacted for future studies will be part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Former Glowing and Expecting study participants aged 5 to 14 years of age

Exclusion Criteria:

* Participants who were dropped from the Glowing and Expecting studies.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Former Glowing and Expecting study participants aged 5 to 14 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 514 (Estimated)
Dates: Start 2017-03-27 (Actual); Primary Completion 2031-03-01 (Estimated); Study Completion 2031-03-01 (Estimated)

PRIMARY OUTCOMES:
Child's growth and development | up to age 14
  Will be determined with body composition equipment (DXA and NMR)
Child's metabolism and physical activity | up to age 14
  Will be determined with metabolic cart and fitness test equipment

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No